CLINICAL TRIAL: NCT06363331
Title: Efficacy of the Social Cognition Rehabilitation Program E-motional Training (ET®) in the Treatment of Patients With Substance-related Disorders and Development of Biomarkers Predicting Response Through Proteomics
Brief Title: Efficacy of the Social Cognition Rehabilitation Program E-motional Training in the Treatment of Patients With Substance-related Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020I054
Record Dates: First submitted 2024-01-31; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-02

CONDITIONS: Social Behavior
Keywords: sustance related disorder
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients TRS without social cognition damage (No Intervention): Patients TRS without damage without intervention
- Patients TRS with Social Cognition control (No Intervention): Patients TRS with social cognition damage with regular therapy in the centre
- Patients TRS with social cognition with Emotional Training (Experimental): Patients TRS with social cognition damage with Emotional Training therapy in the centre
  Interventions: Behavioral: Emotional Training

INTERVENTIONS:
Behavioral: Emotional Training — Emotional Training Therapy following the programme in the computer
  Arms: Patients TRS with social cognition with Emotional Training

SUMMARY:
Drug use, substance use disorders (SUD) and other addictive behaviors are problems of enormous socio-health impact that still require a great research effort to improve the diagnostic and therapeutic procedures used in healthcare practice.

Since addictive behaviors have been consistently associated with the presence of alterations in cognitive and executive functions, it is necessary to be able to detect, evaluate and have specific therapies for these dysfunctions and investigate, among other issues, the role they play in the onset and course evolutionary. After implementing neuropsychological evaluation techniques for diagnostic improvement, addresses the search for procedures that allow working on cognitive and executive deficits, as a specific therapeutic target.

To characterize the presence of alterations in the domains that make up social cognition (SC) in patients with SUD and test in our healthcare units the ET® program already tested both experimentally and at beta level. It is an online self-training program for CS rehabilitation that includes modules for emotion recognition (RE), Theory of Mind (ToM) and attributional style (AS).

To replicate the RCT carried out in schizophrenia in patients with SUD with difficulties in RE or ToM, in addition to searching for a biomarker or a pattern of them that predict the patient profile that will benefit from the training, using advanced LC-ESI proteomics techniques. MS/MS in saliva since previous studies in a population with schizophrenia, subjected to different neurorehabilitation therapies. It is also intended to subsequently improve the instrument (ET®) through the implementation of big data analysis and machine learning and the introduction of automated user management. At this level, the objective is to determine, after the first games, the type of game and the intensity required to improve the user's performance until it reaches normality.

From the perspective of the State Plan for Scientific and Technical Research and Innovation, this project combines CLINICAL AND TRANSLATIONAL RESEARCH, based on the evidence of scientific and technological knowledge, and the use of ENABLING TECHNOLOGIES of e-health in the area of Health Services. Health for people with SUD.

DETAILED DESCRIPTION:
HYPOTHESIS: There is evidence on the existence of social cognition (SC) dysfunctions in patients with SUD and its potential implications in the etiopathogenesis, clinical course and response to treatment have been postulated. At the healthcare level, CS should be taken into account in diagnostic and therapeutic procedures.

The detection of SC dysfunctions and the implementation of specific treatment for them will contribute to improving the therapeutic response of patients with SUD.

GENERAL OBJECTIVES:

1. To study the presence of CS dysfunctions in a clinical sample of patients treated in drug addiction care facilities.
2. To study the therapeutic efficacy of the ET® program in patients with SUD who present SC dysfunctions.
3. Identify new biomarkers in saliva, using mass spectrometry techniques (LC-ESI-MS/MS), that contribute to predicting patients who would benefit from receiving therapy with the ET® program.
4. Improve the ET® instrument to serve new types of users, both in the healthcare and educational environments, and for future adaptation to commercial exploitation.

SPECIFIC OBJECTIVES:

1.1 Evaluate the presence of dysfunctions in the subdomains of the CS 1.2 Evaluate gender differences in the presence of SC dysfunctions 2.1 Evaluate the effectiveness of ET® to improve CS in patients with SUD. 2.2 Evaluate the effectiveness of ET® on the therapeutic response: adherence, quality of life, symptomatological perception, relapses.

2.3 Gender differences in the efficacy of ET® treatment 3.1 Identify molecular patterns in saliva that are associated with SC dysfunctions 3.2 Identify biomarkers that predict therapeutic response. 3.1 Evaluate gender differences in the study of biomarkers 4.1 Collect observations and suggestions from participating researchers to improve the ET® 4.2 Collect observations and suggestions from participating patients for the improvement of the ET®

Methodology (subjects, variables, data collection, analysis plan):

To study the presence of SC dysfunctions in a clinical sample of patients treated in drug addiction care facilities, patients with a diagnosis of SUD who begin treatment in care centers in Galicia, the Valencian Community and Portugal will be recruited to carry out the phase of collecting sociodemographic variables. , descriptive and psychometric evaluation using the battery described below.

To study the therapeutic efficacy of the ET® program in patients with SUD who present SC dysfunctions, a multicenter, longitudinal, prospective, controlled and randomized multimodal (proteomic, neurocognitive and clinical) study phase on the effectiveness of ET® will be carried out. Early prediction of response in patients with SUD requiring social cognition rehabilitation treatment. The response will be evaluated after 3 months (short term), after 12 sessions where activities on emotions and theory of mind are combined, and a follow-up will be carried out after 12 months (long term).

To identify new biomarkers in saliva, using mass spectrometry techniques (LC-ESI-MS/MS), which contribute to predicting patients who would benefit from receiving therapy with the ET® program, saliva samples will be collected to carry out the proteomic study in all participants in the ET® efficacy trial To improve the ET® instrument to serve new types of users, both in the healthcare and educational environment, and for its future adaptation for commercial exploitation, observations and evaluations of researchers and patients will be recorded in order to implement potential future ET® improvements STUDY POPULATION: Patients who begin treatment in care facilities of the drug addiction network, who meet the selection criteria specified in the inclusion criteria section and who do not meet any of the exclusion criteria.

NEUROPSYCHOLOGICAL ASSESSMENT (pre and post):

The neuropsychological evaluation time is estimated at 180 minutes. For the proposed protocol, at least 3 evaluation sessions are required:

* The assessment of cognitive/executive functioning requires a 30-minute session.
* The assessment of social cognition requires 2 sessions of 75 minutes

Patients will be evaluated before and after the intervention, and the evaluation will be repeated after 12 months, using the instruments described below:

Cognitive functioning

* Wechsler Scale for the Measurement of Intelligence in Adults and Adolescents (WAIS III)
* STROOP test
* D2 Attention Test Social cognition
* Innuendo test
* Ekman 60 Faces Test
* Happé's strange stories
* Movie for the Assessment of Social Cognition (MASC)
* Ambiguous Intentions Hostility Questionnaire (AIHQ)

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with substance-related disorders (SUD) and other addictions according to DSM-5 diagnosed by an expert clinician.
* Have the capacity to consent (competence).
* Read the project information sheet and sign the informed consent.
* Age>18 years-old

Exclusion Criteria:

* Illiterate
* Intellectual deficiency defined as IQ<70,
* History of moderate or severe neurological pathology (TBI, stroke, etc.),
* Current acute psychiatric process
* Abstinence of less than 15 days,
* Advanced cognitive impairment that does not allow evaluation.
* Have participated in another similar study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Assess the presence of dysfunctions in the subdomains of social cognition | up to 12 months
  Social cognition by MASC test

SECONDARY OUTCOMES:
Accuracy and efficacy of ET® in patients with SDB | up to 12 months
  Social cognition by AIHQ test

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Galicia Sur Health Research Institute (IISGS) - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Galicia Sur Health Research Institute, Vigo, Pontevedra

IPD SHARING:
Plan to Share IPD: No